CLINICAL TRIAL: NCT06356272
Title: Oropharynx (OPX) Biomarker Trial
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 19-006036; NCI-2024-00965 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-006036 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Metastatic Oropharyngeal Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Head and Neck Carcinoma; Head and Neck Neoplasm; Salivary Gland Neoplasms; Thyroid Gland Neoplasm
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma; Head and Neck Neoplasms; Salivary Gland Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants indicate whether their biospecimen samples (tissue from surgical sample, blood samples, and/or saliva samples) can be retained after the study for future research use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood sample collection, saliva sample collection, complete questionnaires and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
The purpose of this research is to identify a biomarker that is exists when human papillomavirus (HPV) mediated oropharyngeal squamous cell carcinoma is present and does not exist when HPV mediated oropharyngeal squamous cell carcinoma is absent.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify a biomarker (or biomarkers) that is present when disease is present (i.e., at diagnosis or recurrence) and not present when disease is absent (i.e., after treatment, in HPV negative patients or in normal controls).

OUTLINE: This is an observational study.

Patients undergo blood sample collection, saliva sample collection, complete questionnaires and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to provide written consent
* Groups 1-3:

  * Must undergo p16 staining on biopsy for enrollment
  * Patients with < 70% of tumor cells positive for p16 will be considered p16 negative
  * Must undergo HPV16 family in situ hybridization (ISH) and/or RNA on biopsy or surgical specimen, unless amount of tissue is too small to have conclusive HPV ISH testing done on it
  * Willingness and intent to return in person to enrolling institution for follow-up (during the Active Monitoring Phase of the study) for at least 2 of the standard follow-up time points for a total of 3 time-points including pre-treatment. A participant who does not return in person to Mayo Clinic Rochester for every standard of care post-treatment follow up will not be considered deviating from the protocol
* Group 4:

  * Clinical suspicion or histopathologic diagnosis of head and neck cancer or neoplasm

    * Primary salivary neoplasm
    * Primary thyroid neoplasm
    * Primary head and neck neoplasm
    * Multi-cancer early detection (MCED) testing concerning for cancer
* Patient has given permission to give his/her tumor/tissue/blood/saliva sample for research testing
* Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm.
* Groups 1-3:

  * Other active malignancy ≤ 5 years prior to registration

    * EXCEPTIONS: Non-melanotic skin cancer, non-metastatic thyroid cancer, non-metastatic prostate cancer, carcinoma-in-situ of the cervix, HPV+ oropharyngeal squamous cell carcinoma (SCC) (which can be enrolled in group 3)
    * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
  * History of any head and neck malignancy, other than the tumor for which they are being treated
* Group 4, Cohort A, B, C:

  * Other active malignancy ≤ 5 years prior to registration

    * EXCEPTIONS: Non-metastatic prostate cancer, carcinoma-in-situ of the cervix, non metastatic cutaneous basal cell carcinoma
    * NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
  * History of any head and neck malignancy, other than the present neoplasm
  * Note these are clarifications of inclusion into Group 4, Cohorts D and E:

    * Presence of other active malignancy or recurrent head and neck neoplasms are allowed in this arm
    * Receipt of cancer specific therapy for other malignancy is allowed in this arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults > 18 years of age with newly diagnosed untreated, progressive, or metastatic oropharyngeal squamous cell carcinoma with known HPV status
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in biomarkers | Up to 24 months
  Biospecimen samples will be assessed for a biomarker (or biomarkers) that is present when disease is present (i.e., at diagnosis or recurrence) and not present when disease is absent (i.e., after treatment, in HPV negative patients or in normal controls).
Oncologic outcomes associated with biomarkers | Up to study completionUp to 24 months
  Survival outcome (overall survival, disease-free survival, and distant failure) will be compared with blood, tissue and saliva biomarkers identified throughout the treatment course.
Genetic alterations | Up to 24 months
  Alterations in oropharynx tumor specimens will be compared with the detection rate of corresponding circulating DNA in oropharynx cancer patients throughout their treatment course
Immunologic biomarkers for diagnosis | Up to 24 months
  Detected immunologic biomarkers will be compared with overall survival to determine whether biomarkers can be used to predict diagnosis.
Immunologic biomarkers for prognosis | Up to 24 months
  Detected immunologic biomarkers will be compared with overall survival to determine whether biomarkers can be used to predict prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M. Van Abel, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials